CLINICAL TRIAL: NCT02862223
Title: Neprinol for Cardiovascular Health
Brief Title: A Study Investigating the Effects of Neprinol Study Product on Vascular Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KGK Science Inc. (Industry)
Collaborators: Arthur Andrew Medical (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AAME1000
Record Dates: First submitted 2016-07-28; First posted 2016-08-10 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Obesity; Overweight
Keywords: Coagulation; Circulatory Function; Blood Pressure; Inflammatory response; Blood Glucose; Healthy vascular function
MeSH Terms: conditions — Obesity; Overweight; Thrombosis

ARMS (1):
- Neoprinol (Experimental)
  Interventions: Dietary Supplement: Neoprinol

INTERVENTIONS:
Dietary Supplement: Neoprinol

SUMMARY:
This open-label study investigated the effectiveness of Neprinol on maintaining healthy cardiovascular health in overweight and obese adults. Subjects took 3 capsules, 3 times per day over a period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female ≥ 18 and ≤ 75 years of age.
* Overweight subjects (BMI ≥ 27 and < 30) and Obese subjects (BMI > 30 and ≤ 35)
* Subjects with elevated cholesterol.

  * Total cholesterol 240 mg/dL.
* Subjects with elevated inflammation

  * HS-CRP ≥ 3 mg/L.
* Judged by the Investigator to be in general good health on the basis of medical history.
* Females of child bearing potential must agree to use appropriate birth control methods during the entire study period.
* Agree not to initiate any new exercise or diet programs during the entire study period.
* Agree not to change their current diet or exercise program during the entire study period.
* Understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study investigator.

Exclusion Criteria:

* Subjects with a history of congestive heart failure (any classification), unstable angina, or acute coronary syndrome within the past 30 days.
* Uncontrolled hypertension (blood pressure ≥ 170/100 mm Hg)
* Subjects with a history of gastrointestinal disease or surgery affecting absorption
* Subjects with peripheral arterial disease
* Daily use of NSAIDs, however 81mg of aspirin daily for cardio protection is allowed
* Daily use of anti-inflammatory or omega-3-fatty acid dietary supplements

  * 2 week washout is allowed
* Use of any immunosuppressive drugs in the last 12 months (including steroids or biologics)
* Any significant GI condition that would severely interfere with the evaluation of the study product including but not limited to inflammatory bowel disease (Ulcerative Colitis or Chron's), history of frequent diarrhea, history of surgery for weight loss (including gastric bypass or lapband), history of perforation of the stomach or intestines, gastroparesis, clinically important lactose intolerance
* Subjects with a history of using diabetic medications during the prior 4 weeks to study start
* Subjects with a history of using insulin during prior 12 weeks to study start.
* Any active infection, or infection in the last month requiring antibiotics, anti-viral medication, or hospitalization
* History or presence of cancer in the prior two years, except for non-melanoma skin cancer.
* Subjects with a history of seizure
* Recent history of (within 12 months) or strong potential for alcohol or substance abuse.
* Participation in a clinical study with exposure to any non-registered drug product within 30 days prior.
* Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk. Including subjects who are Bed or wheelchair-bound
* Untreated or unstable Hypothyroidism
* Subjects with active eating disorder including anorexia nervosa, bulimia, and/or obsessive compulsive eating disorders
* Pregnant, lactating, or unwilling to use adequate contraception during the duration of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-03; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The change in levels of D-Dimer after 12 weeks of supplementation with the study product. | 12 weeks
The change in levels of Fibrinogen after 12 weeks of supplementation with the study product. | 12 weeks
The change in levels of PAI-1 after 12 weeks of supplementation with the study product. | 12 weeks
The change in levels of Fibrin Monomer after 12 weeks of supplementation with the study product. | 12 weeks
The change in levels of Thrombin anti-thrombin III after 12 weeks of supplementation with the study product. | 12 weeks
The change in levels of ESR after 12 weeks of supplementation with the study product. | 12 weeks
The change in levels of PTT after 12 weeks of supplementation with the study product. | 12 weeks
The change in levels of PT-INR after 12 weeks of supplementation with the study product. | 12 weeks
The change in levels of Activated Clotting Time after 12 weeks of supplementation with the study product. | 12 weeks
The change in levels of Platelet Count after 12 weeks of supplementation with the study product. | 12 weeks
The change in Whole Blood Viscosity after 12 weeks of supplementation with the study | 12 weeks

SECONDARY OUTCOMES:
The change in circulatory function after 12 weeks of supplementation with the study product, measured by EndoPAT analysis | 12 weeks
The change in blood pressure after 12 weeks of supplementation with the study | 12 weeks
The change in levels of HS-CRP after 12 weeks of supplementation with the study product | 12 weeks
The change in levels of Adiponectin after 12 weeks of supplementation with the study product | 12 weeks
The change in levels of IL-6 after 12 weeks of supplementation with the study product | 12 weeks
  Change in inflammatory markers after 12 weeks of supplementation with Neprinol. Inflammatory markers: HS-CRP, Adiponectin, IL-6, TNF-alpha, VEGF
The change in levels of VEGF after 12 weeks of supplementation with the study product | 12 weeks
The change in levels of TNF-alpha after 12 weeks of supplementation with the study product | 12 weeks
The change in NK Cell Cytotoxicity after 12 weeks of supplementation with the study product | 12 weeks
The change in lipid levels after 12 weeks of supplementation with the study product, measured as LDL, HDL and TG | 12 weeks
The change in Glucose AUC after 12 weeks of supplementation with the study product | 12 weeks

OTHER OUTCOMES:
The change in CBC levels after 12 weeks of supplementation with the study product | 12 weeks
The number of Adverse Events reported after 12 weeks of supplementation with the study product | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Gillam, Study Director — Arthur Andrew Medical